CLINICAL TRIAL: NCT03170362
Title: PRIME Care (PRecision Medicine In MEntal Health Care)
Acronym: PRIME Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDR 16-348
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Major Depression
Keywords: Treatment; Pharmacogenetics; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: The study intervention is the provision of pharmacogenetic test results which can then be used to choice appropriate medication.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Pharmacogenetic test results will be provided to the provider within 72 hours of randomization in order to facilitate choice in selecting antidepressants.
  Interventions: Other: Pharmacogenetic Test
- Delay results group (No Intervention): The comparator arm will not receive results at the time of randomization but will get results after the 24 week assessment (thus the results are delayed).

INTERVENTIONS:
Other: Pharmacogenetic Test — The intervention is a battery of pharmacogenetic test results that mostly affect the metabolism of antidepressants and other medications.
  Arms: Intervention group

SUMMARY:
The focus of this application is on the impact of providing depressed Veterans and their providers with the results of pharmacogenetic (PGx) testing for psychotropic medications. The project focuses on whether and how patients and providers use genetic test results given to them at the time an antidepressant is to be initiated to treat Major Depressive Disorder (MDD) and whether use of the test results improves patient outcomes. MDD is one of the most common conditions associated with military service and combat exposure, increases suicide risk, and worsens the course of common medical conditions, making it a leading cause of functional impairment and mortality. Validation of a PGx test to personalize the treatment of MDD represents an important opportunity to improve the healthcare of Veterans.

DETAILED DESCRIPTION:
Background: In the last several years, commercial pharmacogenetic (PGx) testing for psychotropic medications has become widespread as a means of implementing "precision medicine", with some insurers electing to cover the cost of testing. These developments have put increasing pressure on the Veterans Health Administration to implement a mental health focused PGxs program, especially for treating depression, but without sufficient scientific study to support the utility of clinical application.

Objectives: The investigators propose a program of research to evaluate the utility of PGx testing in treating Major Depressive Disorder.

Methods: The investigators plan a multi-site RCT (n=2000), patient/provider dyads will be randomly assigned to receive results of the PGx battery right after randomization (i.e. intervention group) or after 6 months of treatment as usual (i.e. delayed results group)The study will test the following hypotheses:

1. Veterans with MDD whose care is guided by the results of the PGx battery (the intervention group) will have a higher rate of remission of depression than the delayed results group. (Primary Hypothesis)
2. Provider/patient dyads in the intervention group will use fewer medications that have potential gene-drug interactions based on commercial PGx test results than dyads in the delayed results group (Primary Hypothesis).

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 score 10 and a presumptive diagnosis of MDD per PHQ-9 criteria
* at least one prior treatment exposure for MDD (psychotherapy or antidepressant
* intent to start treatment of the MDD with an antidepressant, simple dose increases will not be considered inclusionary
* willingness to provide signed, informed consent to participate in the study

Exclusion Criteria:

* current serious co-occurring psychiatric illness, i.e.:

  * schizophrenia
  * bipolar disorder
  * psychotic major depression
  * borderline or antisocial personality disorder
  * eating disorder
* active alcohol or other drug use disorder
* current use of an antipsychotic medication
* augmentation therapy, e.g.:

  * use of two or more antidepressants at the time of randomization (trazodone at a dosage < 150 mg/day will not be considered augmentation and thus allowed)
* patients requiring urgent care or inpatient hospitalization at the time of consent
* currently incarcerated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1944 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Oslin, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (24):
- United States (24):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Wilmington VA Medical Center, Wilmington, DE, Wilmington, Delaware
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Access to a final data set will be by request only. The investigators will set up a formal approval process which will include a request form. The investigators will require requests to include hypotheses and specify data variables requested. Requests will be reviewed by the Executive Committee for approval. If approved, the requestor will be given a user agreement specifying how the data may be used. Once the agreement is signed and returned, the investigators will provide the requester with an anonymized data set via secure transit method. The investigators will also publish a data dictionary and a primer of our research methods.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 7/1/2022
Access Criteria: published with article

REFERENCES:
- [Background] de Zwarte SMC, Brouwer RM, Agartz I, Alda M, Aleman A, Alpert KI, Bearden CE, Bertolino A, Bois C, Bonvino A, Bramon E, Buimer EEL, Cahn W, Cannon DM, Cannon TD, Caseras X, Castro-Fornieles J, Chen Q, Chung Y, De la Serna E, Di Giorgio A, Doucet GE, Eker MC, Erk S, Fears SC, Foley SF, Frangou S, Frankland A, Fullerton JM, Glahn DC, Goghari VM, Goldman AL, Gonul AS, Gruber O, de Haan L, Hajek T, Hawkins EL, Heinz A, Hillegers MHJ, Hulshoff Pol HE, Hultman CM, Ingvar M, Johansson V, Jonsson EG, Kane F, Kempton MJ, Koenis MMG, Kopecek M, Krabbendam L, Kramer B, Lawrie SM, Lenroot RK, Marcelis M, Marsman JC, Mattay VS, McDonald C, Meyer-Lindenberg A, Michielse S, Mitchell PB, Moreno D, Murray RM, Mwangi B, Najt P, Neilson E, Newport J, van Os J, Overs B, Ozerdem A, Picchioni MM, Richter A, Roberts G, Aydogan AS, Schofield PR, Simsek F, Soares JC, Sugranyes G, Toulopoulou T, Tronchin G, Walter H, Wang L, Weinberger DR, Whalley HC, Yalin N, Andreassen OA, Ching CRK, van Erp TGM, Turner JA, Jahanshad N, Thompson PM, Kahn RS, van Haren NEM. The Association Between Familial Risk and Brain Abnormalities Is Disease Specific: An ENIGMA-Relatives Study of Schizophrenia and Bipolar Disorder. Biol Psychiatry. 2019 Oct 1;86(7):545-556. doi: 10.1016/j.biopsych.2019.03.985. Epub 2019 Jun 13. PMID 31443932
- [Background] Leroux AJ, Waid-Ebbs JK, Wen PS, Helmer DA, Graham DP, O'Connor MK, Ray K. An Investigation of Exposure Control Methods With Variable-Length CAT Using the Partial Credit Model. Appl Psychol Meas. 2019 Nov;43(8):624-638. doi: 10.1177/0146621618824856. Epub 2019 Jan 23. PMID 31551640
- [Background] Sun Y, Chang S, Wang F, Sun H, Ni Z, Yue W, Zhou H, Gelernter J, Malison RT, Kalayasiri R, Wu P, Lu L, Shi J. Genome-wide association study of alcohol dependence in male Han Chinese and cross-ethnic polygenic risk score comparison. Transl Psychiatry. 2019 Oct 7;9(1):249. doi: 10.1038/s41398-019-0586-3. PMID 31591379
- [Background] Nievergelt CM, Maihofer AX, Klengel T, Atkinson EG, Chen CY, Choi KW, Coleman JRI, Dalvie S, Duncan LE, Gelernter J, Levey DF, Logue MW, Polimanti R, Provost AC, Ratanatharathorn A, Stein MB, Torres K, Aiello AE, Almli LM, Amstadter AB, Andersen SB, Andreassen OA, Arbisi PA, Ashley-Koch AE, Austin SB, Avdibegovic E, Babic D, Baekvad-Hansen M, Baker DG, Beckham JC, Bierut LJ, Bisson JI, Boks MP, Bolger EA, Borglum AD, Bradley B, Brashear M, Breen G, Bryant RA, Bustamante AC, Bybjerg-Grauholm J, Calabrese JR, Caldas-de-Almeida JM, Dale AM, Daly MJ, Daskalakis NP, Deckert J, Delahanty DL, Dennis MF, Disner SG, Domschke K, Dzubur-Kulenovic A, Erbes CR, Evans A, Farrer LA, Feeny NC, Flory JD, Forbes D, Franz CE, Galea S, Garrett ME, Gelaye B, Geuze E, Gillespie C, Uka AG, Gordon SD, Guffanti G, Hammamieh R, Harnal S, Hauser MA, Heath AC, Hemmings SMJ, Hougaard DM, Jakovljevic M, Jett M, Johnson EO, Jones I, Jovanovic T, Qin XJ, Junglen AG, Karstoft KI, Kaufman ML, Kessler RC, Khan A, Kimbrel NA, King AP, Koen N, Kranzler HR, Kremen WS, Lawford BR, Lebois LAM, Lewis CE, Linnstaedt SD, Lori A, Lugonja B, Luykx JJ, Lyons MJ, Maples-Keller J, Marmar C, Martin AR, Martin NG, Maurer D, Mavissakalian MR, McFarlane A, McGlinchey RE, McLaughlin KA, McLean SA, McLeay S, Mehta D, Milberg WP, Miller MW, Morey RA, Morris CP, Mors O, Mortensen PB, Neale BM, Nelson EC, Nordentoft M, Norman SB, O'Donnell M, Orcutt HK, Panizzon MS, Peters ES, Peterson AL, Peverill M, Pietrzak RH, Polusny MA, Rice JP, Ripke S, Risbrough VB, Roberts AL, Rothbaum AO, Rothbaum BO, Roy-Byrne P, Ruggiero K, Rung A, Rutten BPF, Saccone NL, Sanchez SE, Schijven D, Seedat S, Seligowski AV, Seng JS, Sheerin CM, Silove D, Smith AK, Smoller JW, Sponheim SR, Stein DJ, Stevens JS, Sumner JA, Teicher MH, Thompson WK, Trapido E, Uddin M, Ursano RJ, van den Heuvel LL, Van Hooff M, Vermetten E, Vinkers CH, Voisey J, Wang Y, Wang Z, Werge T, Williams MA, Williamson DE, Winternitz S, Wolf C, Wolf EJ, Wolff JD, Yehuda R, Young RM, Young KA, Zhao H, Zoellner LA, Liberzon I, Ressler KJ, Haas M, Koenen KC. International meta-analysis of PTSD genome-wide association studies identifies sex- and ancestry-specific genetic risk loci. Nat Commun. 2019 Oct 8;10(1):4558. doi: 10.1038/s41467-019-12576-w. PMID 31594949
- [Background] Cheng Z, Phokaew C, Chou YL, Lai D, Meyers JL, Agrawal A, Farrer LA, Kranzler HR, Gelernter J. A regulatory variant of CHRM3 is associated with cannabis-induced hallucinations in European Americans. Transl Psychiatry. 2019 Nov 18;9(1):309. doi: 10.1038/s41398-019-0639-7. PMID 31740666
- [Background] Wendt FR, Muniz Carvalho C, Pathak GA, Gelernter J, Polimanti R. Deciphering the Biological Mechanisms Underlying the Genome-Wide Associations between Computerized Device Use and Psychiatric Disorders. J Clin Med. 2019 Nov 21;8(12):2040. doi: 10.3390/jcm8122040. PMID 31766499
- [Background] Marees AT, Gamazon ER, Gerring Z, Vorspan F, Fingal J, van den Brink W, Smit DJA, Verweij KJH, Kranzler HR, Sherva R, Farrer L; International Cannabis Consortium; Gelernter J, Derks EM. Post-GWAS analysis of six substance use traits improves the identification and functional interpretation of genetic risk loci. Drug Alcohol Depend. 2020 Jan 1;206:107703. doi: 10.1016/j.drugalcdep.2019.107703. Epub 2019 Nov 4. PMID 31785998
- [Background] Vreeker A, Fears SC, Service SK, Pagani L, Takahashi JS, Araya C, Araya X, Bejarano J, Lopez MC, Montoya G, Montoya CP, Teshiba TM, Escobar J, Cantor RM, Lopez-Jaramillo C, Macaya G, Molina J, Reus VI, Sabatti C, Ophoff RA, Freimer NB, Bearden CE. Genetic analysis of activity, brain and behavioral associations in extended families with heavy genetic loading for bipolar disorder. Psychol Med. 2021 Feb;51(3):494-502. doi: 10.1017/S0033291719003416. Epub 2019 Dec 9. PMID 31813409
- [Background] Hettema JM, Verhulst B, Chatzinakos C, Bacanu SA, Chen CY, Ursano RJ, Kessler RC, Gelernter J, Smoller JW, He F, Jain S, Stein MB. Genome-wide association study of shared liability to anxiety disorders in Army STARRS. Am J Med Genet B Neuropsychiatr Genet. 2020 Jun;183(4):197-207. doi: 10.1002/ajmg.b.32776. Epub 2019 Dec 30. PMID 31886626
- [Background] Levey DF, Gelernter J, Polimanti R, Zhou H, Cheng Z, Aslan M, Quaden R, Concato J, Radhakrishnan K, Bryois J, Sullivan PF; Million Veteran Program; Stein MB. Reproducible Genetic Risk Loci for Anxiety: Results From approximately 200,000 Participants in the Million Veteran Program. Am J Psychiatry. 2020 Mar 1;177(3):223-232. doi: 10.1176/appi.ajp.2019.19030256. Epub 2020 Jan 7. PMID 31906708
- [Background] Cox JW, Sherva RM, Lunetta KL, Johnson EC, Martin NG, Degenhardt L, Agrawal A, Nelson EC, Kranzler HR, Gelernter J, Farrer LA. Genome-Wide Association Study of Opioid Cessation. J Clin Med. 2020 Jan 9;9(1):180. doi: 10.3390/jcm9010180. PMID 31936517
- [Background] Hartwell EE, Feinn R, Morris PE, Gelernter J, Krystal J, Arias AJ, Hoffman M, Petrakis I, Gueorguieva R, Schacht JP, Oslin D, Anton RF, Kranzler HR. Systematic review and meta-analysis of the moderating effect of rs1799971 in OPRM1, the mu-opioid receptor gene, on response to naltrexone treatment of alcohol use disorder. Addiction. 2020 Aug;115(8):1426-1437. doi: 10.1111/add.14975. Epub 2020 Feb 11. PMID 31961981
- [Background] Munn-Chernoff MA, Johnson EC, Chou YL, Coleman JRI, Thornton LM, Walters RK, Yilmaz Z, Baker JH, Hubel C, Gordon S, Medland SE, Watson HJ, Gaspar HA, Bryois J, Hinney A, Leppa VM, Mattheisen M, Ripke S, Yao S, Giusti-Rodriguez P, Hanscombe KB, Adan RAH, Alfredsson L, Ando T, Andreassen OA, Berrettini WH, Boehm I, Boni C, Boraska Perica V, Buehren K, Burghardt R, Cassina M, Cichon S, Clementi M, Cone RD, Courtet P, Crow S, Crowley JJ, Danner UN, Davis OSP, de Zwaan M, Dedoussis G, Degortes D, DeSocio JE, Dick DM, Dikeos D, Dina C, Dmitrzak-Weglarz M, Docampo E, Duncan LE, Egberts K, Ehrlich S, Escaramis G, Esko T, Estivill X, Farmer A, Favaro A, Fernandez-Aranda F, Fichter MM, Fischer K, Focker M, Foretova L, Forstner AJ, Forzan M, Franklin CS, Gallinger S, Giegling I, Giuranna J, Gonidakis F, Gorwood P, Gratacos Mayora M, Guillaume S, Guo Y, Hakonarson H, Hatzikotoulas K, Hauser J, Hebebrand J, Helder SG, Herms S, Herpertz-Dahlmann B, Herzog W, Huckins LM, Hudson JI, Imgart H, Inoko H, Janout V, Jimenez-Murcia S, Julia A, Kalsi G, Kaminska D, Karhunen L, Karwautz A, Kas MJH, Kennedy JL, Keski-Rahkonen A, Kiezebrink K, Kim YR, Klump KL, Knudsen GPS, La Via MC, Le Hellard S, Levitan RD, Li D, Lilenfeld L, Lin BD, Lissowska J, Luykx J, Magistretti PJ, Maj M, Mannik K, Marsal S, Marshall CR, Mattingsdal M, McDevitt S, McGuffin P, Metspalu A, Meulenbelt I, Micali N, Mitchell K, Monteleone AM, Monteleone P, Nacmias B, Navratilova M, Ntalla I, O'Toole JK, Ophoff RA, Padyukov L, Palotie A, Pantel J, Papezova H, Pinto D, Rabionet R, Raevuori A, Ramoz N, Reichborn-Kjennerud T, Ricca V, Ripatti S, Ritschel F, Roberts M, Rotondo A, Rujescu D, Rybakowski F, Santonastaso P, Scherag A, Scherer SW, Schmidt U, Schork NJ, Schosser A, Seitz J, Slachtova L, Slagboom PE, Slof-Op't Landt MCT, Slopien A, Sorbi S, Swiatkowska B, Szatkiewicz JP, Tachmazidou I, Tenconi E, Tortorella A, Tozzi F, Treasure J, Tsitsika A, Tyszkiewicz-Nwafor M, Tziouvas K, van Elburg AA, van Furth EF, Wagner G, Walton E, Widen E, Zeggini E, Zerwas S, Zipfel S, Bergen AW, Boden JM, Brandt H, Crawford S, Halmi KA, Horwood LJ, Johnson C, Kaplan AS, Kaye WH, Mitchell J, Olsen CM, Pearson JF, Pedersen NL, Strober M, Werge T, Whiteman DC, Woodside DB, Grove J, Henders AK, Larsen JT, Parker R, Petersen LV, Jordan J, Kennedy MA, Birgegard A, Lichtenstein P, Norring C, Landen M, Mortensen PB, Polimanti R, McClintick JN, Adkins AE, Aliev F, Bacanu SA, Batzler A, Bertelsen S, Biernacka JM, Bigdeli TB, Chen LS, Clarke TK, Degenhardt F, Docherty AR, Edwards AC, Foo JC, Fox L, Frank J, Hack LM, Hartmann AM, Hartz SM, Heilmann-Heimbach S, Hodgkinson C, Hoffmann P, Hottenga JJ, Konte B, Lahti J, Lahti-Pulkkinen M, Lai D, Ligthart L, Loukola A, Maher BS, Mbarek H, McIntosh AM, McQueen MB, Meyers JL, Milaneschi Y, Palviainen T, Peterson RE, Ryu E, Saccone NL, Salvatore JE, Sanchez-Roige S, Schwandt M, Sherva R, Streit F, Strohmaier J, Thomas N, Wang JC, Webb BT, Wedow R, Wetherill L, Wills AG, Zhou H, Boardman JD, Chen D, Choi DS, Copeland WE, Culverhouse RC, Dahmen N, Degenhardt L, Domingue BW, Frye MA, Gaebel W, Hayward C, Ising M, Keyes M, Kiefer F, Koller G, Kramer J, Kuperman S, Lucae S, Lynskey MT, Maier W, Mann K, Mannisto S, Muller-Myhsok B, Murray AD, Nurnberger JI, Preuss U, Raikkonen K, Reynolds MD, Ridinger M, Scherbaum N, Schuckit MA, Soyka M, Treutlein J, Witt SH, Wodarz N, Zill P, Adkins DE, Boomsma DI, Bierut LJ, Brown SA, Bucholz KK, Costello EJ, de Wit H, Diazgranados N, Eriksson JG, Farrer LA, Foroud TM, Gillespie NA, Goate AM, Goldman D, Grucza RA, Hancock DB, Harris KM, Hesselbrock V, Hewitt JK, Hopfer CJ, Iacono WG, Johnson EO, Karpyak VM, Kendler KS, Kranzler HR, Krauter K, Lind PA, McGue M, MacKillop J, Madden PAF, Maes HH, Magnusson PKE, Nelson EC, Nothen MM, Palmer AA, Penninx BWJH, Porjesz B, Rice JP, Rietschel M, Riley BP, Rose RJ, Shen PH, Silberg J, Stallings MC, Tarter RE, Vanyukov MM, Vrieze S, Wall TL, Whitfield JB, Zhao H, Neale BM, Wade TD, Heath AC, Montgomery GW, Martin NG, Sullivan PF, Kaprio J, Breen G, Gelernter J, Edenberg HJ, Bulik CM, Agrawal A. Shared genetic risk between eating disorder- and substance-use-related phenotypes: Evidence from genome-wide association studies. Addict Biol. 2021 Jan;26(1):e12880. doi: 10.1111/adb.12880. Epub 2020 Feb 16. PMID 32064741
- [Background] Dalvie S, Maihofer AX, Coleman JRI, Bradley B, Breen G, Brick LA, Chen CY, Choi KW, Duncan LE, Guffanti G, Haas M, Harnal S, Liberzon I, Nugent NR, Provost AC, Ressler KJ, Torres K, Amstadter AB, Bryn Austin S, Baker DG, Bolger EA, Bryant RA, Calabrese JR, Delahanty DL, Farrer LA, Feeny NC, Flory JD, Forbes D, Galea S, Gautam A, Gelernter J, Hammamieh R, Jett M, Junglen AG, Kaufman ML, Kessler RC, Khan A, Kranzler HR, Lebois LAM, Marmar C, Mavissakalian MR, McFarlane A, Donnell MO, Orcutt HK, Pietrzak RH, Risbrough VB, Roberts AL, Rothbaum AO, Roy-Byrne P, Ruggiero K, Seligowski AV, Sheerin CM, Silove D, Smoller JW, Stein MB, Teicher MH, Ursano RJ, Van Hooff M, Winternitz S, Wolff JD, Yehuda R, Zhao H, Zoellner LA, Stein DJ, Koenen KC, Nievergelt CM. Genomic influences on self-reported childhood maltreatment. Transl Psychiatry. 2020 Jan 27;10(1):38. doi: 10.1038/s41398-020-0706-0. PMID 32066696
- [Background] Polimanti R, Walters RK, Johnson EC, McClintick JN, Adkins AE, Adkins DE, Bacanu SA, Bierut LJ, Bigdeli TB, Brown S, Bucholz KK, Copeland WE, Costello EJ, Degenhardt L, Farrer LA, Foroud TM, Fox L, Goate AM, Grucza R, Hack LM, Hancock DB, Hartz SM, Heath AC, Hewitt JK, Hopfer CJ, Johnson EO, Kendler KS, Kranzler HR, Krauter K, Lai D, Madden PAF, Martin NG, Maes HH, Nelson EC, Peterson RE, Porjesz B, Riley BP, Saccone N, Stallings M, Wall TL, Webb BT, Wetherill L; Psychiatric Genomics Consortium Substance Use Disorders Workgroup; Edenberg HJ, Agrawal A, Gelernter J. Leveraging genome-wide data to investigate differences between opioid use vs. opioid dependence in 41,176 individuals from the Psychiatric Genomics Consortium. Mol Psychiatry. 2020 Aug;25(8):1673-1687. doi: 10.1038/s41380-020-0677-9. Epub 2020 Feb 26. PMID 32099098
- [Background] de Araujo CM, Hudziak J, Crocetti D, Wymbs NF, Montalvo-Ortiz JL, Orr C, Albaugh MD, Althoff RR, O'Loughlin K, Holbrook H, Garavan H, Yang BZ, Mostofsky S, Jackowski A, Lee RS, Gelernter J, Kaufman J. Tubulin Polymerization Promoting Protein (TPPP) gene methylation and corpus callosum measures in maltreated children. Psychiatry Res Neuroimaging. 2020 Apr 30;298:111058. doi: 10.1016/j.pscychresns.2020.111058. Epub 2020 Feb 22. PMID 32120304
- [Background] Muniz Carvalho C, Wendt FR, Maihofer AX, Stein DJ, Stein MB, Sumner JA, Hemmings SMJ, Nievergelt CM, Koenen KC, Gelernter J, Belangero SI, Polimanti R. Dissecting the genetic association of C-reactive protein with PTSD, traumatic events, and social support. Neuropsychopharmacology. 2021 May;46(6):1071-1077. doi: 10.1038/s41386-020-0655-6. Epub 2020 Mar 16. PMID 32179874
- [Background] Hunter-Zinck H, Shi Y, Li M, Gorman BR, Ji SG, Sun N, Webster T, Liem A, Hsieh P, Devineni P, Karnam P, Gong X, Radhakrishnan L, Schmidt J, Assimes TL, Huang J, Pan C, Humphries D, Brophy M, Moser J, Muralidhar S, Huang GD, Przygodzki R, Concato J, Gaziano JM, Gelernter J, O'Donnell CJ, Hauser ER, Zhao H, O'Leary TJ; VA Million Veteran Program; Tsao PS, Pyarajan S. Genotyping Array Design and Data Quality Control in the Million Veteran Program. Am J Hum Genet. 2020 Apr 2;106(4):535-548. doi: 10.1016/j.ajhg.2020.03.004. PMID 32243820
- [Background] Zhou H, Sealock JM, Sanchez-Roige S, Clarke TK, Levey DF, Cheng Z, Li B, Polimanti R, Kember RL, Smith RV, Thygesen JH, Morgan MY, Atkinson SR, Thursz MR, Nyegaard M, Mattheisen M, Borglum AD, Johnson EC, Justice AC, Palmer AA, McQuillin A, Davis LK, Edenberg HJ, Agrawal A, Kranzler HR, Gelernter J. Genome-wide meta-analysis of problematic alcohol use in 435,563 individuals yields insights into biology and relationships with other traits. Nat Neurosci. 2020 Jul;23(7):809-818. doi: 10.1038/s41593-020-0643-5. Epub 2020 May 25. PMID 32451486
- [Background] Zhou H, Rentsch CT, Cheng Z, Kember RL, Nunez YZ, Sherva RM, Tate JP, Dao C, Xu K, Polimanti R, Farrer LA, Justice AC, Kranzler HR, Gelernter J; Veterans Affairs Million Veteran Program. Association of OPRM1 Functional Coding Variant With Opioid Use Disorder: A Genome-Wide Association Study. JAMA Psychiatry. 2020 Oct 1;77(10):1072-1080. doi: 10.1001/jamapsychiatry.2020.1206. PMID 32492095
- [Background] Wendt FR, Carvalho CM, Pathak GA, Gelernter J, Polimanti R. Polygenic risk for autism spectrum disorder associates with anger recognition in a neurodevelopment-focused phenome-wide scan of unaffected youths from a population-based cohort. PLoS Genet. 2020 Sep 17;16(9):e1009036. doi: 10.1371/journal.pgen.1009036. eCollection 2020 Sep. PMID 32941431
- [Background] McIntyre RS, Subramaniapillai M, Lee Y, Pan Z, Carmona NE, Shekotikhina M, Rosenblat JD, Brietzke E, Soczynska JK, Cosgrove VE, Miller S, Fischer EG, Kramer NE, Dunlap K, Suppes T, Mansur RB. Efficacy of Adjunctive Infliximab vs Placebo in the Treatment of Adults With Bipolar I/II Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Aug 1;76(8):783-790. doi: 10.1001/jamapsychiatry.2019.0779. PMID 31066887
- [Background] Kramer NE, Cosgrove VE, Dunlap K, Subramaniapillai M, McIntyre RS, Suppes T. A clinical model for identifying an inflammatory phenotype in mood disorders. J Psychiatr Res. 2019 Jun;113:148-158. doi: 10.1016/j.jpsychires.2019.02.005. Epub 2019 Feb 10. PMID 30954775
- [Background] Ward RE, Cho K, Nguyen XT, Vassy JL, Ho YL, Quaden RM, Gagnon DR, Wilson PWF, Gaziano JM, Djousse L; VA Million Veteran Program. Omega-3 supplement use, fish intake, and risk of non-fatal coronary artery disease and ischemic stroke in the Million Veteran Program. Clin Nutr. 2020 Feb;39(2):574-579. doi: 10.1016/j.clnu.2019.03.005. Epub 2019 Mar 13. PMID 30914216
- [Background] Raghavan S, Vassy JL, Ho YL, Song RJ, Gagnon DR, Cho K, Wilson PWF, Phillips LS. Diabetes Mellitus-Related All-Cause and Cardiovascular Mortality in a National Cohort of Adults. J Am Heart Assoc. 2019 Feb 19;8(4):e011295. doi: 10.1161/JAHA.118.011295. PMID 30776949
- [Background] Hidalgo-Mazzei D, Berk M, Cipriani A, Cleare AJ, Florio AD, Dietch D, Geddes JR, Goodwin GM, Grunze H, Hayes JF, Jones I, Kasper S, Macritchie K, McAllister-Williams RH, Morriss R, Nayrouz S, Pappa S, Soares JC, Smith DJ, Suppes T, Talbot P, Vieta E, Watson S, Yatham LN, Young AH, Stokes PRA. Treatment-resistant and multi-therapy-resistant criteria for bipolar depression: consensus definition. Br J Psychiatry. 2019 Jan;214(1):27-35. doi: 10.1192/bjp.2018.257. Epub 2018 Dec 6. PMID 30520709
- [Background] van der Markt A, Klumpers UM, Draisma S, Dols A, Nolen WA, Post RM, Altshuler LL, Frye MA, Grunze H, Keck PE Jr, McElroy SL, Suppes T, Beekman AT, Kupka RW. Testing a clinical staging model for bipolar disorder using longitudinal life chart data. Bipolar Disord. 2019 May;21(3):228-234. doi: 10.1111/bdi.12727. Epub 2018 Dec 12. PMID 30447123
- [Background] Imran TF, Posner D, Honerlaw J, Vassy JL, Song RJ, Ho YL, Kittner SJ, Liao KP, Cai T, O'Donnell CJ, Djousse L, Gagnon DR, Gaziano JM, Wilson PW, Cho K. A phenotyping algorithm to identify acute ischemic stroke accurately from a national biobank: the Million Veteran Program. Clin Epidemiol. 2018 Oct 16;10:1509-1521. doi: 10.2147/CLEP.S160764. eCollection 2018. PMID 30425582
- [Background] Post RM, Altshuler LL, Kupka R, McElroy SL, Frye MA, Rowe M, Grunze H, Suppes T, Keck PE Jr, Leverich GS, Nolen WA. Multigenerational transmission of liability to psychiatric illness in offspring of parents with bipolar disorder. Bipolar Disord. 2018 Jun 21. doi: 10.1111/bdi.12668. Online ahead of print. PMID 29926532
- [Background] Nielsen DA, Spellicy CJ, Harding MJ, Graham DP. Apolipoprotein E DNA methylation and posttraumatic stress disorder are associated with plasma ApoE level: A preliminary study. Behav Brain Res. 2019 Jan 1;356:415-422. doi: 10.1016/j.bbr.2018.05.013. Epub 2018 May 26. PMID 29807071
- [Background] Yatham LN, Kennedy SH, Parikh SV, Schaffer A, Bond DJ, Frey BN, Sharma V, Goldstein BI, Rej S, Beaulieu S, Alda M, MacQueen G, Milev RV, Ravindran A, O'Donovan C, McIntosh D, Lam RW, Vazquez G, Kapczinski F, McIntyre RS, Kozicky J, Kanba S, Lafer B, Suppes T, Calabrese JR, Vieta E, Malhi G, Post RM, Berk M. Canadian Network for Mood and Anxiety Treatments (CANMAT) and International Society for Bipolar Disorders (ISBD) 2018 guidelines for the management of patients with bipolar disorder. Bipolar Disord. 2018 Mar;20(2):97-170. doi: 10.1111/bdi.12609. Epub 2018 Mar 14. PMID 29536616
- [Background] Vieta E, Berk M, Schulze TG, Carvalho AF, Suppes T, Calabrese JR, Gao K, Miskowiak KW, Grande I. Bipolar disorders. Nat Rev Dis Primers. 2018 Mar 8;4:18008. doi: 10.1038/nrdp.2018.8. PMID 29516993
- [Background] Gonzalez R, Suppes T, Zeitzer J, McClung C, Tamminga C, Tohen M, Forero A, Dwivedi A, Alvarado A. The association between mood state and chronobiological characteristics in bipolar I disorder: a naturalistic, variable cluster analysis-based study. Int J Bipolar Disord. 2018 Feb 19;6(1):5. doi: 10.1186/s40345-017-0113-5. PMID 29457195
- [Background] Post RM, Leverich GS, McElroy S, Kupka R, Suppes T, Altshuler L, Nolen W, Frye M, Keck P, Grunze H, Hellemann G. Prevalence of axis II comorbidities in bipolar disorder: relationship to mood state. Bipolar Disord. 2018 Jun;20(4):303-312. doi: 10.1111/bdi.12596. Epub 2018 Jan 25. PMID 29369448
- [Background] Williams LM, Pines A, Goldstein-Piekarski AN, Rosas LG, Kullar M, Sacchet MD, Gevaert O, Bailenson J, Lavori PW, Dagum P, Wandell B, Correa C, Greenleaf W, Suppes T, Perry LM, Smyth JM, Lewis MA, Venditti EM, Snowden M, Simmons JM, Ma J. The ENGAGE study: Integrating neuroimaging, virtual reality and smartphone sensing to understand self-regulation for managing depression and obesity in a precision medicine model. Behav Res Ther. 2018 Feb;101:58-70. doi: 10.1016/j.brat.2017.09.012. Epub 2017 Oct 7. PMID 29074231
- [Background] Lippard ETC, Jensen KP, Wang F, Johnston JAY, Spencer L, Pittman B, Gelernter J, Blumberg HP. Genetic variation of ANK3 is associated with lower white matter structural integrity in bipolar disorder. Mol Psychiatry. 2017 Sep;22(9):1225. doi: 10.1038/mp.2017.169. No abstract available. PMID 28831200
- [Background] Stein MB, Chen CY, Jain S, Jensen KP, He F, Heeringa SG, Kessler RC, Maihofer A, Nock MK, Ripke S, Sun X, Thomas ML, Ursano RJ, Smoller JW, Gelernter J; Army STARRS Collaborators. Genetic risk variants for social anxiety. Am J Med Genet B Neuropsychiatr Genet. 2017 Jun;174(4):470-482. doi: 10.1002/ajmg.b.32541. Epub 2017 Apr 27. No abstract available. PMID 28512750
- [Background] Stein MB, Chen CY, Jain S, Jensen KP, He F, Heeringa SG, Kessler RC, Maihofer A, Nock MK, Ripke S, Sun X, Thomas ML, Ursano RJ, Smoller JW, Gelernter J; Army STARRS Collaborators. Genetic risk variants for social anxiety. Am J Med Genet B Neuropsychiatr Genet. 2017 Mar;174(2):120-131. doi: 10.1002/ajmg.b.32520. PMID 28224735
- [Background] Polimanti R, Zhang H, Smith AH, Zhao H, Farrer LA, Kranzler HR, Gelernter J. Genome-wide association study of body mass index in subjects with alcohol dependence. Addict Biol. 2017 Mar;22(2):535-549. doi: 10.1111/adb.12317. Epub 2015 Oct 12. PMID 26458734
- [Result] Hull LE, Lynch KG, Oslin DW. VA Primary Care and Mental Health Providers' Comfort with Genetic Testing: Survey Results from the PRIME Care Study. J Gen Intern Med. 2019 Jun;34(6):799-801. doi: 10.1007/s11606-018-4776-0. No abstract available. PMID 30604117
- [Result] Chanfreau-Coffinier C, Hull LE, Lynch JA, DuVall SL, Damrauer SM, Cunningham FE, Voight BF, Matheny ME, Oslin DW, Icardi MS, Tuteja S. Projected Prevalence of Actionable Pharmacogenetic Variants and Level A Drugs Prescribed Among US Veterans Health Administration Pharmacy Users. JAMA Netw Open. 2019 Jun 5;2(6):e195345. doi: 10.1001/jamanetworkopen.2019.5345. PMID 31173123
- [Result] Hull LE, Chanfreau-Coffinier C, Tuteja S, Berlowitz D, Lehmann LS, Oslin DW, Pyne JM, DuVall SL, Lynch JA. Early adoption of pharmacogenetic testing for veterans prescribed psychotropic medications. Pharmacogenomics. 2019 Jul;20(11):781-789. doi: 10.2217/pgs-2019-0065. Epub 2019 Aug 8. PMID 31393222
- [Result] Oslin DW, Chapman S, Duvall SL, Gelernter J, Ingram EP, Kranzler HR, Lehmann LS, Lynch JA, Lynch KG, Pyne JM, Shih MC, Stone A, Thase ME, Wray LO. Study design and implementation of the PRecision Medicine In MEntal health Care (PRIME Care) Trial. Contemp Clin Trials. 2021 Feb;101:106247. doi: 10.1016/j.cct.2020.106247. Epub 2020 Dec 11. PMID 33316457
- [Result] Vest BM, Wray LO, Brady LA, Thase ME, Beehler GP, Chapman SR, Hull LE, Oslin DW. Primary care and mental health providers' perceptions of implementation of pharmacogenetics testing for depression prescribing. BMC Psychiatry. 2020 Oct 28;20(1):518. doi: 10.1186/s12888-020-02919-z. PMID 33115428
- [Result] Ramsey CM, Lynch KG, Thase ME, Gelernter J, Kranzler HR, Pyne JM, Shih MC, Stone A; PRIME Care Executive Committee; Oslin DW. Prevalence of predicted gene-drug interactions for antidepressants in the treatment of major depressive disorder in the Precision Medicine in Mental Health Care Study. J Affect Disord. 2021 Mar 1;282:1272-1277. doi: 10.1016/j.jad.2021.01.034. Epub 2021 Jan 14. PMID 33601706
- [Result] Oslin DW, Lynch KG, Shih MC, Ingram EP, Wray LO, Chapman SR, Kranzler HR, Gelernter J, Pyne JM, Stone A, DuVall SL, Lehmann LS, Thase ME; PRIME Care Research Group; Aslam M, Batki SL, Bjork JM, Blow FC, Brenner LA, Chen P, Desai S, Dieperink EW, Fears SC, Fuller MA, Goodman CS, Graham DP, Haas GL, Hamner MB, Helstrom AW, Hurley RA, Icardi MS, Jurjus GJ, Kilbourne AM, Kreyenbuhl J, Lache DJ, Lieske SP, Lynch JA, Meyer LJ, Montalvo C, Muralidhar S, Ostacher MJ, Paschall GY, Pfeiffer PN, Prieto S, Przygodzki RM, Ranganathan M, Rodriguez-Suarez MM, Roggenkamp H, Schichman SA, Schneeweis JS, Simonetti JA, Steinhauer SR, Suppes T, Umbert MA, Vassy JL, Voora D, Wiechers IR, Wood AE. Effect of Pharmacogenomic Testing for Drug-Gene Interactions on Medication Selection and Remission of Symptoms in Major Depressive Disorder: The PRIME Care Randomized Clinical Trial. JAMA. 2022 Jul 12;328(2):151-161. doi: 10.1001/jama.2022.9805. PMID 35819423
- [Result] Ziobrowski HN, Cui R, Ross EL, Liu H, Puac-Polanco V, Turner B, Leung LB, Bossarte RM, Bryant C, Pigeon WR, Oslin DW, Post EP, Zaslavsky AM, Zubizarreta JR, Nierenberg AA, Luedtke A, Kennedy CJ, Kessler RC. Development of a model to predict psychotherapy response for depression among Veterans. Psychol Med. 2023 Jun;53(8):3591-3600. doi: 10.1017/S0033291722000228. Epub 2022 Feb 11. PMID 35144713
- [Result] Na PJ, De Angelis F, Nichter B, Wendt FR, Krystal JH, Southwick SM, Levey DF, Gelernter J, Polimanti R, Pietrzak RH. Psychosocial moderators of polygenic risk for suicidal ideation: Results from a 7-year population-based, prospective cohort study of U.S. veterans. Mol Psychiatry. 2022 Feb;27(2):1068-1074. doi: 10.1038/s41380-021-01352-2. Epub 2021 Nov 2. PMID 34725455
- [Result] Tamman AJF, Wendt FR, Pathak GA, Krystal JH, Southwick SM, Sippel LM, Gelernter J, Polimanti R, Pietrzak RH. Attachment Style Moderates Polygenic Risk for Incident Posttraumatic Stress in U.S. Military Veterans: A 7-Year, Nationally Representative, Prospective Cohort Study. Biol Psychiatry. 2022 Apr 1;91(7):637-646. doi: 10.1016/j.biopsych.2021.09.025. Epub 2021 Oct 6. PMID 34955171
- [Result] Montalvo-Ortiz JL, Gelernter J, Cheng Z, Girgenti MJ, Xu K, Zhang X, Gopalan S, Zhou H, Duman RS, Southwick SM, Krystal JH; Traumatic Stress Brain Research Study Group; Pietrzak RH. Epigenome-wide association study of posttraumatic stress disorder identifies novel loci in U.S. military veterans. Transl Psychiatry. 2022 Feb 17;12(1):65. doi: 10.1038/s41398-022-01822-3. PMID 35177594
- [Result] Verma A, Huffman JE, Gao L, Minnier J, Wu WC, Cho K, Ho YL, Gorman BR, Pyarajan S, Rajeevan N, Garcon H, Joseph J, McGeary JE, Suzuki A, Reaven PD, Wan ES, Lynch JA, Petersen JM, Meigs JB, Freiberg MS, Gatsby E, Lynch KE, Zekavat SM, Natarajan P, Dalal S, Jhala DN, Arjomandi M, Bonomo RA, Thompson TK, Pathak GA, Zhou JJ, Donskey CJ, Madduri RK, Wells QS, Gelernter J, Huang RDL, Polimanti R, Chang KM, Liao KP, Tsao PS, Sun YV, Wilson PWF, O'Donnell CJ, Hung AM, Gaziano JM, Hauger RL, Iyengar SK, Luoh SW; VA Million Veteran Program COVID-19 Science Initiative. Association of Kidney Comorbidities and Acute Kidney Failure With Unfavorable Outcomes After COVID-19 in Individuals With the Sickle Cell Trait. JAMA Intern Med. 2022 Aug 1;182(8):796-804. doi: 10.1001/jamainternmed.2022.2141. PMID 35759254
- [Result] Na PJ, Montalvo-Ortiz JL, Nagamatsu ST, Southwick SM, Krystal JH, Gelernter J, Pietrzak RH. Association of Symptoms of Posttraumatic Stress Disorder and GrimAge, an Epigenetic Marker of Mortality Risk, in US Military Veterans. J Clin Psychiatry. 2022 Jul 6;83(4):21br14309. doi: 10.4088/JCP.21br14309. No abstract available. PMID 35802930
- [Derived] Reis DJ, Kinney AR, Forster JE, Stearns-Yoder KA, Kittel JA, Wood AE, Oslin DW, Brenner LA, Simonetti JA. Longitudinal invariance of the Patient Health Questionnaire-9 among patients receiving pharmacotherapy for major depressive disorder: A secondary analysis of clinical trial data. Psychol Assess. 2024 Aug;36(8):462-471. doi: 10.1037/pas0001317. Epub 2024 May 16. PMID 38753374
- [Derived] Chanfreau-Coffinier C, Tuteja S, Hull LE, MacDonald S, Efimova O, Bates J, Voora D, Oslin DW, DuVall SL, Lynch JA. Drug-drug-gene interaction risk among opioid users in the U.S. Department of Veterans Affairs. Pain. 2022 Dec 1;163(12):2390-2397. doi: 10.1097/j.pain.0000000000002637. Epub 2022 Mar 23. PMID 35319502
- [Derived] Ramsey CM, Lynch KG, Gehrman PR, Vairavan S, Narayan VA, Li QS, Oslin DW. Daily steps and depressive symptoms: A longitudinal evaluation of patients with major depressive disorder in the precision medicine in mental health care study. J Affect Disord. 2022 Mar 1;300:334-340. doi: 10.1016/j.jad.2021.12.116. Epub 2022 Jan 1. PMID 34979178
- See also: Website location for educational materials — https://www.mirecc.va.gov/visn4/PrimeCare/PRIME_Care.asp

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Delay Results Group
Started | 966 | 978
Completed | 754 | 787
Not Completed | 212 | 191
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 23 | 22
Not completed — Lost to Follow-up | 187 | 167

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Delay Results Group | Total
Number analyzed (Participants) | 966 | 978 | 1944
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (15) | 47 (15) | 48 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 262 | 491
  Male | 737 | 716 | 1453
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 113 | 104 | 217
  Not Hispanic or Latino | 850 | 869 | 1719
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 9 | 19
  Asian | 31 | 24 | 55
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 185 | 167 | 352
  White | 644 | 688 | 1332
  More than one race | 90 | 84 | 174
  Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 966 | 978 | 1944
Depression severity [Mean (Standard Deviation); unit: units on a scale] — PHQ9 assessment measures depression severity. Min = 0 Max=27, higher scores indicate greater severity.
  units on a scale | 17.5 (4.3) | 17.5 (4.3) | 17.5 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Depression Remission
Description: The investigators will use the Patient Health Questionnaire 9 (PHQ9) as a self assessed marker of depression remission. The scale ranges from 0 to 27 with lower scores indicating less depression severity. Remission was defined as a score of 5 or less at the endpoint. the reported number of participants are those reaching that threshold of symptoms.
Time Frame: 24 weeks post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Delay Results Group
Number analyzed (Participants) | 754 | 787
Participants | 130 | 126

2. Primary Outcome: Use of Fewer Medications That Have Potential Gene-drug Interactions
Description: The investigators will examine the proportion of antidepressants prescribed in the first 30 days of the trial that have the potential for gene-drug interactions. The chance for a gene-drug interaction was classified as 1. the subject did not have a prescription for an antidepressant during the initial 4 weeks of the trial (No Antidepressant), 2 the subject was prescribed an antidepressant with no known gene-drug interaction (No Gene Interaction), 3 the subject was prescribed an antidepressant with moderate gene-drug interactions (Moderate Interaction). These are also gene-drug interactions that do not have level A concordance. And 4. the subject was prescribed an antidepressant with substantial gene-drug interactions or gene-drug interactions that are considered to have a high level of evidence to support other prescribing.
Time Frame: Over the first 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Delay Results Group
Number analyzed (Participants) | 966 | 978
Participants
  No Antidepressant prescibed | 239 | 299
  Taking an antidepressant with no gene interaction | 433 | 173
  Taking an antidepressant with moderate gene interaction | 215 | 373
  Taking an antidepressant with substantial gene interaction | 79 | 133

3. Secondary Outcome: Depression Severity
Description: The investigators will use the Patient Health Questionnaire 9 (PHQ9) as a self-assessed marker of depression remission. The scale ranges from 0 to 27 with lower scores indicating less depression severity. This measure will use the PHQ9 as a continuous measure. The reported outcome is the difference in scores from baseline to 24 weeks.
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Delay Results Group
Number analyzed (Participants) | 754 | 787
units on a scale | 5.4 (5.9) | 4.8 (5.6)

4. Secondary Outcome: Depression Response
Description: The investigators will use the Patient Health Questionnaire 9 (PHQ9) as a self assessed marker of depression remission. The scale ranges from 0 to 27 with lower scores indicating less depression severity. Response was measured by a 50% reduction in scores from baseline to each time point.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Delay Results Group
Number analyzed (Participants) | 754 | 787
Participants | 242 | 216

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Intervention Group | Delay Results Group
All-Cause Mortality (participants affected / at risk) | 2/966 | 2/978
Serious Adverse Events (participants affected / at risk) | 76/966 | 70/978
Other Adverse Events (participants affected / at risk) | 650/966 | 636/978
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=966) | Delay Results Group (N=978)
Hospitalization (Cardiac disorders) | 11 (11) | 8 (9)
Hospitalization (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Hospitalization (Endocrine disorders) | 3 (6) | 2 (2)
Hospitalization (Gastrointestinal disorders) | 8 (10) | 12 (13)
Hospitalization (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hospitalization (Infections and infestations) | 8 (8) | 6 (8)
Hospitalization (Nervous system disorders) | 6 (6) | 7 (7)
Hospitalization (Psychiatric disorders) | 18 (24) | 18 (24)
Incarceration (Social circumstances) | 0 (0) | 1 (1)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (7)
Hospitalization (Renal and urinary disorders) | 1 (1) | 2 (2)
Hospitalization (Musculoskeletal and connective tissue disorders) | 13 (13) | 7 (8)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=966) | Delay Results Group (N=978)
Headache (Nervous system disorders) | 345 (676) | 370 (705)
Sexual side effects (Reproductive system and breast disorders) | 409 (982) | 402 (1026)
GI distress (Gastrointestinal disorders) | 272 (461) | 235 (417)
Nausea (Gastrointestinal disorders) | 272 (461) | 235 (417)
Fatigue (Nervous system disorders) | 130 (185) | 108 (161)
Insomnia (Nervous system disorders) | 54 (64) | 62 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT03170362/Prot_002.pdf
  • Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT03170362/SAP_000.pdf
  • Informed Consent Form (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT03170362/ICF_001.pdf